CLINICAL TRIAL: NCT06540820
Title: NEUROENDOCRINE REGULATION OF BONE-FAT CROSSTALK IN OBESITY
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Federico II University (Other); University of Catanzaro (Other); Istituto Auxologico Italiano (Other)
Responsible Party: Principal Investigator, Andrea Giustina, Professor, IRCCS San Raffaele
Other Study IDs: PNRR-MCNT1-2023-12377758
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Obesity; Endocrine; Pituitary Dysfunction; Bone Health
MeSH Terms: conditions — Obesity | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with pituitary disorders
  Interventions: Diagnostic Test: Dexa or Biompedance analysis with clinical and biochemical evaluations
- patients without pituitary disorders
  Interventions: Diagnostic Test: Dexa or Biompedance analysis with clinical and biochemical evaluations

INTERVENTIONS:
Diagnostic Test: Dexa or Biompedance analysis with clinical and biochemical evaluations — All patients will undergo body composition study with DXA or Bioimpedance analysis which are the gold standard to determine % of fat mass and fat free mass, basal biochemical examinations and oral glucose tolerance test (OGTT), and clinical evaluation with waist circumference measurement. Moreover, all patients will undergo REMS ultrasound, TBS and BSI evaluation at DXA scan and hand grip test. In addition, all patients will undergo to clinical evaluation with specific nutritional, physical activity and sleep quality questionnaire assessments and an additional volume of blood.

SUMMARY:
To study the effect of neuroendocrine dysfunctions on bone health in obesity

DETAILED DESCRIPTION:
It is a multicentric, observational, cross-sectional non-profit study with additional procedures. The study will include obese patients (BMI>30) with and without hyper functioning pituitary adenomas (acromegaly, Cushing and prolactinoma) and hypopituitarism (GH deficiency, secondary hypogonadism) aimed at studying the effect of metabolic phenotypes of obesity and neuroendocrine dysfunctions on bone health.

Patients enrollment will take place in Ospedale San Raffaele, Azienda Ospedaliera Universitaria Federico II di Napoli and UOC Endocrinologia-AOU Renato Dulbecco, Università degli Studi di Catanzaro Magna Graecia.

ELIGIBILITY:
Inclusion criteria for subjects with pituitary disease:

* Male and female subject > 18-year-old (also fertile patients can be included)
* Patients with prolactinoma or Cushing disease, Acromegaly or hypogonadism/hypopituitarism
* BMI ≥30 Kg/m2
* Able to sign an informed consent

Inclusion criteria for subjects without pituitary disease

* Male and female subject > 18-year-old
* BMI ≥ 30 Kg/m2
* Able to sign an informed consent

Exclusion Criteria:

* Male and female subject <18-year-old
* pregnant or breastfeeding women
* Subject unable to sign informed consent
* BMI < 30 Kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients with or without pituitary/gonadal disorders will be enrolled. Patients enrollment will take place in Ospedale San Raffaele, Azienda Ospedaliera Universitaria Federico II di Napoli and UOC Endocrinologia-AOU Renato Dulbecco, Università degli Studi di Catanzaro Magna Graecia.
  A total of n=150 obese individuals will be recruited as it follows:
  1. n=30 obese patients with acromegaly
  2. n=30 obese patients with hyperprolactinemia
  3. n=30 obese patients with hypopituitarism, including secondary male hypogonadism
  4. n=30 obese patients with Cushing syndrome
  5. n=30 obese patients without neuroendocrine diseases as control group
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
To study the neuroendocrine control of bone-fat crosstalk in obesity. Obese patients with and without neuroendocrine dysfunctions will be enrolled in the study to evaluate bone health, as well as the content of circulating adipokines/osteokines. | 2 weeks
  The following assessments will be performed:
  1. Biochemical exams to determine the presence of primary or secondary hypogonadism or other alterations of the neuroendocrine axis.
  2. Bone health: -Blood and urine samples -Hip, lumbar and ultradistal BMD by DXA; -Vertebral fractures assessment on lateral dorso-lumbar spine DXA scans by a quantitative morphometric approach. -Bone microarchitectural and microstructural characteristics, performing TBS. -Distal HRpQCT -Bone Strain index (BSi) parameters from hip and lumbar DXA scans, obtaining a qualitative index of bone strength based on finite element analysis.
  b) Adipokines and obesity-associated cytokines serum content. c) Osteokines serum content.

IPD SHARING:
Plan to Share IPD: No